CLINICAL TRIAL: NCT03686644
Title: Effects of Wearing Orthoses on Nightly Postures on Passive Stiffness in Plantar Flexors Muscles in Children With Cerebral Palsy
Brief Title: Ankle-foot Orthoses for Night Splinting in Children With CP: Impact on Passive Stiffness in Plantarflexors Muscles
Acronym: NIGHTSTRETCH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: never started
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18CH070; 2018-A01082-53 (Other: ANSM)
Record Dates: First submitted 2018-09-24; First posted 2018-09-27 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Cerebral Palsy
Keywords: night splinting; stiffness; ankle foot orthoses; teenager
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with Cerebral Palsy (Experimental): Children with Cerebral Palsy (CP) will be included. They will have to wearing of night splint ankle foot orthoses (phase A) and then no wearing of night splint ankle foot orthoses (phase B). The phases A and B will be repeated twice. In more, they will have an ultrasound, isokinetic dynamometer and measure of quality of night sleeping.
  Interventions: Procedure: Wearing of night splint ankle foot orthoses (phase A); Procedure: No wearing of night splint ankle foot orthoses (phase B)

INTERVENTIONS:
Procedure: Wearing of night splint ankle foot orthoses (phase A) — Children wearing of night splint ankle foot orthoses during 6, 7 or 8 days according to the position of inclusion.
  An ultrasound of the leg muscles will be realized every morning after removing night splint.
  An isokinetic dynamometer will be realize at the beginning of the study and at the end of each phase.
  measure of quality of night sleeping will be measured by Visual Analog Scale (VAS) results.
Procedure: No wearing of night splint ankle foot orthoses (phase B) — Children no wearing of night splint ankle foot orthoses during 6, 7 or 8 days according to the position of inclusion.
  An ultrasound of the leg muscles will be realized every morning after removing night splint.
  An isokinetic dynamometer will be realize at the beginning of the study and at the end of each phase.
  measure of quality of night sleeping will be measured by Visual Analog Scale (VAS) results.

SUMMARY:
Children with cerebral palsy present early in the childhood altered muscular properties, characterized by short muscle belly length and increased stiffness which contribute to contracture and limiting joint range of motion. In order to prevent equinus deformity, ankle foot orthoses for night splinting are usually used in children with spastic Cerebral Palsy (CP). However, there's a lack of proof about efficacy by using this modality of treatment. Moreover, impact on quality of life for children and families, cost for society were high.

Principal purpose of this study was to assess impact of night splint ankle foot orthoses on passive stiffness in plantarflexors muscles in children with CP.

DETAILED DESCRIPTION:
Children with cerebral palsy present early in the childhood altered muscular properties, characterized by short muscle belly length and increased stiffness which contribute to contracture and limiting joint range of motion. In order to prevent equinus deformity, ankle foot orthoses for night splinting are usually used in children with spastic CP. However, there's a lack of proof about efficacy by using this modality of treatment. Moreover, impact on quality of life for children and families, cost for society were high.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed spastic cerebral palsy
* Children wearing night splint ankle foot orthoses all night long during 1 week minimum
* Children with a level of spasticity in the gastrocnemius muscle greater than or equal to X1, VII, on the Tardieu scale and 2 on the Ashworth scale.
* Children able to understand and respect the simple instructions of the study
* Children and parents who received informed information about the study and who co-signed, with the investigator, a consent to participate in the study.

Exclusion Criteria:

* Children who do not tolerate ankle foot orthoses all night long.
* Children who had botulinum injection in gastrocnemius or soleus muscles during last three months.
* Children benefiting from an injection of botulinum toxin or the setting up of new equipment during the protocol.
* Children who do not tolerate ankle foot orthoses all night long.
* Children having benefited from plaster lengthening for less than three months.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
change from baseline elasticity modulus of the leg muscles at 4 weeks | Weeks 0, 1, 2, 3 and 4
  measured by ultrasounds

SECONDARY OUTCOMES:
Maximal dorsiflexion angle | Weeks 0, 1, 2, 3 and 4
  Measured by isokinetic dynamometer.
Maximum angle of tense knee dorsiflexion | Weeks 0, 1, 2, 3 and 4
  Measured by isokinetic dynamometer.
Torque of force maximal tolerated in maximum angle of tense knee dorsiflexion | Weeks 0, 1, 2, 3 and 4
  Measured by isokinetic dynamometer.
Visual Analog Scale of sleeping | Weeks 0, 1, 2, 3 and 4
  Measured the quality of night sleeping between 0 (bad sleeping) and 10 (good sleeping).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GAUTHERON, MD PhD, Principal Investigator — CHU de Saint Etienne

IPD SHARING:
Plan to Share IPD: No